CLINICAL TRIAL: NCT04582838
Title: Photoplethysmographic Signal Analysis as a Proxy for Excessive Effort and Impending Respiratory Failure
Brief Title: Photoplethysmographic Scaling of Dyspnoea
Acronym: DYSPO
Status: Completed | Type: Observational
Sponsor: Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu (Other)
Responsible Party: Principal Investigator, Balan Ion Cosmin, Consultant in Anaesthesia and ICM, Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu
Other Study IDs: 18751; Dyspnoea - SpO2 curve study (Other: CC Iliescu Institute)
Record Dates: First submitted 2020-10-04; First posted 2020-10-12 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Respiratory Failure
Keywords: breathing; effort; plethysmography; pulse oximetry; dyspnoea; mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration; Dyspnea | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spontaneous breathing ICU non-COVID: Spontaneously breathing non-COVID-19 critically ill patients with sinus rhythm.
  Inclusion and exclusion criterion are listed elsewhere.
  Interventions: Diagnostic Test: Pulse oximeter; Diagnostic Test: ECG
- Spontaneous breathing ICU COVID: Spontaneously breathing COVID-19 critically ill patients with sinus rhythm.
  Inclusion and exclusion criterion are listed elsewhere.
  Interventions: Diagnostic Test: Pulse oximeter; Diagnostic Test: ECG

INTERVENTIONS:
Diagnostic Test: Pulse oximeter — In both groups, pulse oximeters provide continuous monitoring of oxygen saturation (SpO2).
  Also, SpO2 curve can be recorded for off-line analysis.
Diagnostic Test: ECG — ECG signal is used to monitor respiratory rate (RR).

SUMMARY:
Timely prediction of impending respiratory failure is vital, yet relies on subjective clinical assessment of the patient's respiratory status. Pulse oximetry plethysmographic signal analysis is indicative of the effort to breathe and may provide an objective measurement of respiratory loading.

DETAILED DESCRIPTION:
Initiating invasive mechanical ventilation is a vital and delay-critical decision. Precise and timely prediction of impending respiratory failure would be highly consequential. Subjective evaluation of respiratory loading conditions is inconsistent, imprecise and may result in erroneous management. Photoplethysmographic (POP) waveform analysis provides a non-invasive, readily available tool to estimate breathing effort in a semiquantitative fashion.

It is the aim of this study to examine:

1. if the degree of dyspnoea, when clinically assessed by means of the respiratory rate and SpO2 values, correlates with the SpO2 wave variations (ΔPOP) in ICU spontaneously breathing COVID-19 and non-COVID-19 patients.
2. if a ΔPOP threshold could be identified to adequately predict further need of orotracheal intubation and invasive mechanical ventilation.

This study consists of three main steps:

1. Clinical evaluation of dyspnoea based on:

   1.1. Respiratory rate

   1.2. Oxygen saturation (SpO2)
2. Storage of SpO2 curve for ΔPOP computation according to a proprietary algorithm after offline POP analysis .
3. Within a time frame of 10 days from when the first two steps are met, monitor for need of invasive ventilatory support.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from patient or next-of-kin according to local administrative decision
* Spontaneous breathing, including during prone position
* Sinus rhythm
* Minimum standards for ICU monitoring: ECG, blood pressure (invasive or non-invasive), respiratory rate (by ECG signal), SpO2 and temperature

Exclusion Criteria:

* Suspected pregnancy
* Weight > 120 Kg or < 60 kg
* Emergency or urgency
* Intubated ( and mechanically ventilated) patient
* Non- sinus rhythm
* Left ventricular ejection fraction (LVEF) ≤ 30%
* Right ventricular (RV) dysfunction ( RVEF ≤ 30% at transthoracic echocardiography (TTE))
* Significant pulmonary hypertension (PHT) (TTE: mean pulmonary arterial pressure (mPAP) ≥ 35 mm.Hg)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spontaneously breathing ICU (COVID and non-COVID-19) adult patients with sinus rhythm, under any form of non-invasive respiratory support.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Rate of failure of spontaneous breathing | Day 10
  Number of patients who fail spontaneous breathing (SB). Failure of SB is defined as death or need of invasive mechanical ventilation whereas SB includes any form of non-invasive ventilatory support

SECONDARY OUTCOMES:
Respiratory rate | Day 0
  Patient's respiratory rate during non-invasive respiratory support as derived from an ECG signal
SpO2 under non-invasive respiratory support | Day 0
  Peripheral oxygen saturation (SpO2) as measured with a pulse oximeter during any form of non-invasive ventilatory support
ΔPOP | day 0
  Photoplethysmographic variation index following offline computation of the SpO2 curve stored at day 0 according to a proprietary algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Serban I Bubenek Turconi, Professor, Study Chair — Emergency Institute for Cardiovascular Diseases Prof Dr CC Iliescu
Locations (2):
- Romania (2):
  - Clinical Emergency Hospital Bucharest, Bucharest
  - Clinical Hospital of Infectious and Tropical Diseases "Dr. Victor Babes", Bucharest

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Addison PS. Respiratory effort from the photoplethysmogram. Med Eng Phys. 2017 Mar;41:9-18. doi: 10.1016/j.medengphy.2016.12.010. Epub 2017 Jan 23. PMID 28126420
- [Background] Perel A. Excessive variations in the plethysmographic waveform during spontaneous ventilation: an important sign of upper airway obstruction. Anesth Analg. 2014 Dec;119(6):1288-92. doi: 10.1213/ANE.0000000000000378. PMID 25405690
- [Background] Khandoker AH, Karmakar CK, Penzel T, Glos M, Schoebel C, Palaniswami M. Estimating relative respiratory effort from features of Photo-Plethysmography signal. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:6575-8. doi: 10.1109/EMBC.2013.6611062. PMID 24111249
- [Background] Addison PS. Respiratory modulations in the photoplethysmogram (DPOP) as a measure of respiratory effort. J Clin Monit Comput. 2016 Oct;30(5):595-602. doi: 10.1007/s10877-015-9763-y. Epub 2015 Sep 16. PMID 26377021